CLINICAL TRIAL: NCT00360347
Title: Open Label, Randomized, Exploratory Study to Investigate the Hemoglobin Dose-response, the Safety and the Pharmacokinetic Profile Following Subcutaneous Administration of Mircera Once Every Three Weeks to Anemic Patients With Multiple Myeloma
Brief Title: A Study of Mircera in Anemic Patients With Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA16558
Record Dates: First submitted 2006-08-03; First posted 2006-08-04 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: FDA-regulated Device: No

INTERVENTIONS:
Drug: C.E.R.A.

SUMMARY:
This study will investigate the efficacy, safety and pharmacokinetics of Mircera in adult anemic patients with multiple myeloma. In the first stage of the study, patients will be randomized to receive subcutaneous injections of Mircera once every 3 weeks, at doses of 2.0, 3.5 or 5.0 micrograms/kg. Following the administration of 2 doses, an evaluation of hemoglobin increase will be made at week 6. In the second stage, further groups of patients will receive additional doses of Mircera,at doses of 1.0, 6.5 or 8.0 micrograms/kg, depending on efficacy, safety and pharmacokinetic considerations.The anticipated time on treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* confirmed diagnosis of multiple myeloma;
* anemia (hemoglobin <=11g/dL at screening visit).

Exclusion Criteria:

* transfusion of red blood cells during 2 months prior to first planned dose of study medication;
* therapy-resistant hypertension;
* relevant acute or chronic bleeding within 3 months prior to planned start of study treatment;
* recombinant human erythropoietin or erythropoiesis-stimulating drug therapy within 3 months prior to planned start of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11-29 (Actual); Primary Completion 2003-04-29 (Actual); Study Completion 2003-04-29 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level, and change from baseline, at week 6

SECONDARY OUTCOMES:
Efficacy: Hematocrit, and change from baseline; reticulocyte count. PK:AUC at weeks 4-6; Safety: AEs, laboratory parameters, blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Rokicka, Dr, Principal Investigator — unaffliated
Locations (5):
- Prague, Czechia
- Poland (4):
  - Bialystok
  - Gdansk
  - Lublin
  - Warsaw